CLINICAL TRIAL: NCT02298816
Title: B-Cell Hematologic Malignancy Vaccination Registry
Acronym: HMvax-Regist
Status: Withdrawn | Type: Observational
Why Stopped: No patients enrolled
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Vince Lombardi Cancer Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: HMvax-registry:14-98E
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2024-03

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance; Multiple Myeloma; Waldenstrom Macroglobulinemia; Lymphocytosis; Lymphoma, Non-Hodgkin; B-Cell Chronic Lymphocytic Leukemia; Hematological Malignancies
Keywords: Monoclonal gammopathy of undetermined significance (MGUS); Smoldering multiple myeloma (SMM); Multiple myeloma (MM); Waldenstroms Macroglobulinemia (WM); Monoclonal B-cell lymphocytosis (MBL); Chronic lymphocytic leukemia (CLL); B-Cell Non-Hodgkin lymphoma (NHL); B-Cell Hematologic Malignancies; immunization; Vaccination; Influenza, Human; Pneumonia
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Multiple Myeloma; Waldenstrom Macroglobulinemia; Lymphocytosis; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Hematologic Neoplasms; Smoldering Multiple Myeloma; Lymphoma, B-Cell; Influenza, Human; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- new B-Cell Hematologic Malignancy diagnosis: All adult patients who are newly diagnosed at Aurora Health Care with the following B-Cell Hematologic Malignancies: Monoclonal gammopathy of undetermined significance (MGUS), Smoldering multiple myeloma (SMM), Multiple myeloma (MM), Waldenstroms Macroglobulinemia (WM), Monoclonal B-cell lymphocytosis (MBL), Chronic lymphocytic leukemia (CLL), or B-Cell Non-Hodgkin lymphoma (NHL).

SUMMARY:
The goal of this study is to develop a vaccination registry system for Aurora Health Care patients newly diagnosed with MM and other B-Cell Hematologic Malignancies in order to prospectively characterize vaccination history and outcomes such as infection in these patients at Aurora Health Care. Additionally hospitalization rates, cost analysis, infection (influenza, pneumonia, other) related to vaccination in this patient population will be evaluated.

DETAILED DESCRIPTION:
This is a prospective registry study on the immunizations in patients with B-Cell Hematologic Malignancies at Aurora Health Care. This observational study will consist of prospective medical record review of Aurora Health Care patients newly diagnosed B-Cell Hematologic Malignancies and will be used to characterize vaccination history, infection rate, and hospitalization rate. This is the second study in the series of studies designed to provide important information about the best way and time to vaccinate patients with MM and similar cancers to flu and pneumonia and to gather additional information about immune function in this patient population.

The registry will include all adult patients who are newly diagnosed with the following B-Cell Hematologic Malignancies: Monoclonal gammopathy of undetermined significance (MGUS), Smoldering multiple myeloma (SMM), Multiple myeloma (MM), Waldenstroms Macroglobulinemia (WM), Monoclonal B-cell lymphocytosis (MBL), Chronic lymphocytic leukemia (CLL), or B-Cell Non-Hodgkin lymphoma (NHL). The prevalence of newly diagnosed B-Cell Hematologic Malignancies at Aurora Health Care is approximately 1000 patients annually. This registry will be ongoing to collect real time data, with no definite sample size planned; however, data will be collected for at least 10 years. This time frame is based on Surveillance, Epidemiology, and End Results Program (SEER) data. There is a 50% survival rate at 5 years after diagnosis for MM, so the 10 year time frame will be able to capture long term outcome in patients.

Medical record information will be obtained through electronic data capture by Aurora Health Care staff with access to the electronic medical records. Data will be manually reviewed by the coordinator, Investigator and co-investigators for accuracy and completeness, to the extent available in the clinical medical record. Additionally, a biostatistician will assist in data analysis.

Descriptive statistics such as counts, proportions or percentages for category variables and mean and standard deviation for continuous variables will be computed for the all the variables. Depending upon the distribution of the category variables appropriate statistical tests such as chi-square and/or Fisher exact test will be used to find out the statistical significance. For continuous variables an appropriate statistical test such as t-tests and/or F test will be used.

This registry will be used for this research study, and may be queried for internal quality improvement projects as well. The principal investigator will be responsible for the overall monitoring of the data and safety of study participants/data integrity, with the assistance of other study team members.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at Aurora Health Care who are newly diagnosed with:

  * Monoclonal gammopathy of undetermined significance (MGUS),
  * Smoldering multiple myeloma (SMM),
  * Multiple myeloma (MM),
  * Waldenstroms Macroglobulinemia (WM),
  * Monoclonal B-cell lymphocytosis (MBL),
  * Chronic lymphocytic leukemia (CLL), or
  * B-Cell Non-Hodgkin lymphoma (NHL).

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients at Aurora Health Care who are newly diagnosed with:
  * Monoclonal gammopathy of undetermined significance (MGUS),
  * Smoldering multiple myeloma (SMM),
  * Multiple myeloma (MM),
  * Waldenstroms Macroglobulinemia (WM),
  * Monoclonal B-cell lymphocytosis (MBL),
  * Chronic lymphocytic leukemia (CLL), or
  * B-Cell Non-Hodgkin lymphoma (NHL).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
vaccination history | 10 years
  Information regarding vaccination history will be collected historically and throughout data collection, expected to continue for about 10 years.

SECONDARY OUTCOMES:
Survival | 10 years
  Survival status will be collected throughout data collection, expected to continue for about 10 years.
infection | 10 years
  Information about any infections (influenza, pneumonia, other) such as numbers, types will be collected throughout data collection, expected to continue for about 10 years.
hospitalization rates | 10 years
  Information regarding hospitalization will be collected throughout data collection, expected to continue for about 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thompson, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora Health Care, Milwaukee, Wisconsin, United States